CLINICAL TRIAL: NCT04319263
Title: Oncological Outcomes of Different Patterns of Tumor Recurrence at First Evaluation After Bacillus Calmette-Guérin Induction Therapy for Intermediate and High Risk Non Muscle Invasive Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Principal Investigator, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AE 20320
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intermediate and high risk non muscle invasive bladder cancer (Experimental)
  Interventions: Drug: induction regimen of intravesical BCG

INTERVENTIONS:
Drug: induction regimen of intravesical BCG — intravesical instillation of 6 weekly doses of BCG

SUMMARY:
This retrospective study aimed at assessment of different patterns (morphological and pathological) of tumor recurrence found at first evaluation after BCG induction therapy (3 months cystoscopy) for intermediate and high-risk NMIBC and its prognostic implications at a tertiary referral center.

DETAILED DESCRIPTION:
Bladder cancer (BCa) is the second most common genitourinary malignancy with approximately 75-85% of all patients with BCa present at diagnosis a non-muscle invasive bladder cancer (NMIBC) (Ta, T1 and Tis). Although NMIBC usually carries a favorable prognosis, there is a high risk of disease recurrence and a 10% to 20% risk of progression to muscle-invasive disease.

The common treatment for intermediate- and high-risk patients is a transurethral resection followed by intravesical therapy with bacillus Calmette-Guerin (BCG), a non-specific immunotherapy that has remained the gold standard for 40 years. Over the last decades, several studies have confirmed the superiority of BCG over the combination of epirubicin and interferon, mitomycin C or epirubicin alone for prevention of tumor recurrence, in intermediate- and high-risk tumors.

Despite wide acceptance of BCG intravesical therapy in intermediate and high risk NMIBC, there is still a controversy regarding the optimal protocol of administration. However, most of the guidelines have recommended an induction regimen of six weekly BCG instillations followed by maintenance instillation for at least 1 year.

Complete response (CR) rates after an induction course of BCG for intermediate and high risk NMIBC are high and range from 50-70%. Tumor recurrence at first evaluation (3-months cystoscopy) after BCG induction therapy has been defined as a poor prognostic indicator in those groups of patients with an increased potential risk of disease recurrence and /or progression.

Different patterns of tumor recurrence may be encountered at 3-mo cystoscopy during first evaluation after induction therapy either morphological (single tumor vs. multiple, <3 cm or more, site (? bladder neck involvement), papillary or non papillary) or histopathological (Ta vs. T1, concurrent CIS or not, tumor grade). To determine how to optimally manage those heterogeneous groups of patients, studying of the specific impact of different tumor characteristics on oncological outcomes is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Patients for who complete TURBT, was carried out
* Intermediate and high risk NMIBC.
* Patients who received full induction BCG regimen (6 weekly doses).
* Patients completed at least 12 months follow up after 3 months cystoscopy.

Exclusion Criteria:

* Patients who received incomplete induction BCG regimen (less than 6 weekly doses)
* Patients with incomplete (less than 12 months) follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
one year Recurrence rate | one year
  recurrence rate at 1 year after induction BCG
one year progression rate | one year
  progression rate at 1 year after induction BCG

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Elsawy, Principal Investigator — Urology and Nephrology Center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided